CLINICAL TRIAL: NCT05709860
Title: Adaptation and Pilot Test of an Electronic Health Record-based Approach to Increase PrEP Knowledge and Uptake: the EMC2 PrEP Strategy
Brief Title: An Electronic Health Record-based Approach to Increase PrEP Knowledge and Uptake: the EMC2 PrEP Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Allison Prickett Pack, Research Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00217596
Record Dates: First submitted 2023-01-17; First posted 2023-02-02 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections; Electronic Health Record; Primary Health Care
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care includes: 1) no specific materials to promote PrEP knowledge or uptake among women in primary care, and 2) variable physician counseling on PrEP among women with increased vulnerability to HIV.
- The EMC2 PrEP Strategy (Active Comparator): The EMC2 PrEP Strategy will utilize health information and consumer technologies to automatically deposit an interactive PrEP educational material into the patient portal of women with clinically indicated increased vulnerability to HIV. The material will: 1) promote PrEP knowledge, and 2) prompt discrete scheduling of a dedicated PrEP visit among those interested.
  Interventions: Behavioral: EMC2 PrEP Educational Tool; Behavioral: Discrete Scheduling of a Dedicated PrEP Visit

INTERVENTIONS:
Behavioral: EMC2 PrEP Educational Tool — Patients will receive an interactive PrEP Educational Tool. This interactive tool will be securely sent via the patient portal. After logging into their portal, patients will have the opportunity to review the information on their own time.
  Arms: The EMC2 PrEP Strategy
Behavioral: Discrete Scheduling of a Dedicated PrEP Visit — Within the interactive PrEP Educational Tool, patients who choose to will have the opportunity to discretely schedule a dedicated PrEP visit with a primary care clinician trained on PrEP delivery. The clinician will have time reserved to allow for 'rapid' scheduling.
  Arms: The EMC2 PrEP Strategy

SUMMARY:
This study is being conducted to investigate a strategy that may improve knowledge and uptake of pre-exposure prophylaxis for HIV prevention (PrEP) among cisgender women in primary care.

DETAILED DESCRIPTION:
Members of the study team previously developed and evaluated the Electronic health record Medication Complete Communication (EMC2) strategy to 'hardwire' provider/patient communication & surveillance of select prescription (Rx) medications. EMC2 PrEP will adapt from the previous strategy to

* educate cisgender women in primary care who have increased vulnerability to HIV about PrEP using an interactive, health literacy-appropriate educational tool securely delivered via the patient portal
* facilitate, for those who express interest, the rapid and discrete scheduling of a dedicated PrEP clinic visit with a primary care clinician trained in PrEP delivery

The current study aims are to:

Aim 1: Refine and implement an electronic health record (EHR)-based strategy as a potential quality improvement activity that supports informed decision-making and PrEP uptake among women with increased HIV vulnerability in primary care (the EMC2 PrEP strategy).

Aim 2: Pilot-test the EMC2 PrEP strategy in primary care to determine its feasibility, acceptability, and preliminary efficacy among women with increased vulnerability to HIV.

Aim 3: Develop a standard operating protocol (SOP) for disseminating the EMC2 PrEP strategy to a national network of federally qualified health centers.

ELIGIBILITY:
Inclusion Criteria:

* female
* HIV negative
* have received 2 or more tests in the past 12 months for chlamydia, gonorrhea and/or syphilis
* and/or have received a positive diagnosis for at least one of those sexually transmitted infections in the past 6 months
* currently engaged in primary care
* not currently using PrEP

Exclusion Criteria:

* severe, uncorrectable visual, hearing or cognitive impairments that would preclude study consent or participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Pack, PhD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pack A, O'Conor R, Vasiloff R, Liebovitz D, Masters MC, Alcantara K, Smith R, Wismer G, Tatz R, Yeh F, Curtis LM, Hur S, Bailey SC. An electronic health record-based strategy to increase PrEP decision-making among cisgender women in primary care: results of a randomized pilot study. BMC Health Serv Res. 2025 Apr 24;25(1):589. doi: 10.1186/s12913-025-12745-2. PMID 40269861

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | The EMC2 PrEP Strategy
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | The EMC2 PrEP Strategy | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (9.3) | 36.3 (11.2) | 36.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 14 | 31
  Not Hispanic or Latino | 83 | 86 | 169
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 44 | 45 | 89
  Race: Black/African American | 31 | 35 | 66
  Race: Asian | 8 | 6 | 14
  Race: Other | 10 | 13 | 23
  Race: Multiple | 7 | 1 | 8
Marital Status [Count of Participants; unit: Participants]
  Married | 26 | 32 | 58
  Widowed | 2 | 0 | 2
  Divorced | 9 | 7 | 16
  Separated | 1 | 5 | 6
  Single | 51 | 45 | 96
  Living with a partner | 11 | 7 | 18
  Other | 0 | 4 | 4
Household Income [Count of Participants; unit: Participants] — Population: 1 participant in the intervention group has missing income data.
  Participants
    number analyzed (Participants) | 100 | 99 | 199
    < $25,000 | 7 | 3 | 10
    $25,000-$49,999 | 16 | 14 | 30
    $50,000-$74,999 | 20 | 21 | 41
    $75,000-$99,999 | 13 | 12 | 25
    $100,000 or more | 44 | 49 | 93
Insurance Status [Count of Participants; unit: Participants]
  Private or HMO | 75 | 79 | 154
  Medicaid | 11 | 4 | 15
  Medicare | 2 | 2 | 4
  Self-pay/No insurance | 2 | 1 | 3
  Other | 5 | 7 | 12
  Multiple | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: PrEP Uptake (Use)
Description: PrEP uptake will be measured during the intervention period between study arms to investigate the effects of the EMC2 PrEP strategy.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | The EMC2 PrEP Strategy
Number analyzed (Participants) | 100 | 100
Participants | 0 | 0

2. Secondary Outcome: PrEP Knowledge
Description: A 10-item questionnaire, developed by the study team and the scientific literature, will be used to evaluate knowledge of pre-exposure prophylaxis among study participants. Correctly answered questions will be summed (0 to 10) for a total score. Higher scores will indicate greater PrEP knowledge.
Time Frame: 2-6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | The EMC2 PrEP Strategy
Number analyzed (Participants) | 100 | 100
score on a scale | 5.6 (2.2) | 7.5 (2.5)

3. Secondary Outcome: Perceived Risk of HIV
Description: The 8-item Perceived Risk of HIV scale is used to assess how vulnerable an individual feels to HIV. The scale was developed in the United States and attention was paid to health literacy. Response options vary for each item, though they are measured on a 4-point Likert scale. Total score of 8 items is calculated and range from 10 to 40. Higher scores mean higher perceived risk of HIV.
Time Frame: 2-6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | The EMC2 PrEP Strategy
Number analyzed (Participants) | 100 | 100
score on a scale | 19.2 (5.2) | 19.1 (4.6)

4. Secondary Outcome: PrEP Attitudes
Description: A PrEP Attitudes 5-items scale (Walsh, 2019) is used to assess attitudes toward PrEP, each item is measured on a 5-point Likert scale (1=strongly disagree to 5=strongly agree). A total score is calculated and range from 5 to 25. Higher scores mean more stigma towards PrEP use.
Time Frame: 2-6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | The EMC2 PrEP Strategy
Number analyzed (Participants) | 100 | 100
score on a scale | 11.2 (4.4) | 10.5 (3.9)

5. Secondary Outcome: Health Literacy
Description: CHEW health literacy is used to assess participant's health literacy level. Participants were asked three questions about difficulty in understanding medical materials and information, the options range from all of the time to none of the time. The responses of the three questions are then categorized into limited and adequate health literacy level. We used CHEW health literacy because the measure can be conducted over phone calls.
Time Frame: 2-6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | The EMC2 PrEP Strategy
Number analyzed (Participants) | 100 | 100
Participants
  Limited | 22 | 20
  Adequate | 78 | 80

6. Secondary Outcome: Health Activation
Description: A modified version of our team's 10-item Consumer Health Activation Index (CHAI) is used to assess participant's engagement in healthcare. Response options are a Likert scale; linear transformation is used to put total scores onto a 0-100 scale, with higher numbers indicating greater activation. The total scores are then categorized into 3 categories: Low (0-79), Moderate (80-94), and High (>94).
Time Frame: 2-6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | The EMC2 PrEP Strategy
Number analyzed (Participants) | 100 | 100
Participants
  Low | 61 | 64
  Moderate | 30 | 30
  High | 9 | 6

7. Secondary Outcome: Process Measure
Description: The participants in the intervention group were asked two questions about 1) whether they received a PrEP decision guide, and 2) did they read or review it, to assess the acceptability of the intervention material.
Time Frame: 2-6 weeks
Population: Only participants in the intervention group were asked the questions. 43 participants have missing process measure data.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | The EMC2 PrEP Strategy
Number analyzed (Participants) | 0 | 57
Participants
  Received PrEP decision guide in patient portal |  | 20
  Reviewed the material after received: number analyzed (Participants) | 0 | 20
  Reviewed the material after received |  | 10

8. Secondary Outcome: Acceptability of the Strategy
Description: Using 10-point Likert scale response options (1=very unsatisfied to 10=very satisfied), participants in the intervention group are asked to rate their satisfaction with the materials.
Time Frame: 2-6 weeks
Population: Only the participants in the intervention group are asked to rate their satisfaction with the intervention materials. And 10 participants in the intervention group who read or view the material were asked about the satisfaction with the material.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | The EMC2 PrEP Strategy
Number analyzed (Participants) | 0 | 10
score on a scale
  Satisfaction of the appearance of the guide |  | 7.7 (1.7)
  Satisfaction of the quality of the guide |  | 8.3 (1.8)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed. These were 1-time interviews.
Arm/Group | Usual Care | The EMC2 PrEP Strategy
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT05709860/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT05709860/ICF_001.pdf